CLINICAL TRIAL: NCT04971889
Title: Diabetes Medical Nutrition Therapy in Southeastern African American Women
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meharry Medical College (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Matthew Walker Comprehensive Health Center (Unknown); Vanderbilt University (Other)
Responsible Party: Principal Investigator, Stephania T. Miller-Hughes, Professor, Meharry Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-02-1069
Record Dates: First submitted 2021-07-13; First posted 2021-07-22 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetes MNT plus MI (Active Comparator): --Group-based dietary/dietary motivation intervention
  Interventions: Behavioral: Diabetes MNT; Behavioral: Motivational Interviewing
- Diabetes MNT (Active Comparator): -Group-based dietary intervention
  Interventions: Behavioral: Diabetes MNT

INTERVENTIONS:
Behavioral: Diabetes MNT — Group-based MNT sessions that provide evidence-based dietary self-care information, behavioral skills, and goal setting related to managing carbohydrate and fat intake
Behavioral: Motivational Interviewing — Group-based support for dietary self-care motivation using culturally-adapted motivational interviewing exercise
  Arms: Diabetes MNT plus MI

SUMMARY:
A two-arm randomized controlled trial design will be used. Participants will include 291 African American women with type 2 diabetes that are at risk for development and/or progression of diabetes complications. Both arms, diabetes medical nutrition therapy (MNT) and diabetes MNT plus motivational interviewing (MI), will include: 1) a 3-month active intervention period of six biweekly (every other week), group-based, trained nutritionist-facilitated sessions; 2) a 3-month maintenance intervention period, which will include one group-based maintenance support session; and 3) a 6-month inactive period (no contact). The differences between arms is the integration of culturally-adapted MI exercises during the diabetes MNT plus MI active and maintenance intervention periods.

ELIGIBILITY:
Inclusion Criteria:

* African American
* Female
* Clinical diagnosis of type 2 diabetes for at least 6 months
* At risk for development and/or progression of diabetes complications (HbA1c ≥ 7.0% AND either systolic blood pressure ≥130, LDL cholesterol ≥ 100, or BMI ≥ 30).

Exclusion Criteria:

--Observed or diagnosed psychotic disorders

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identification
Enrollment: 291 (Estimated)
Dates: Start 2021-08-03 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
HbA1c | Baseline
  Widely-utilized high performance liquid chromatography methods will be used to measure glycemic control from whole blood samples.
Change from Baseline HbA1c | 3 months
  Widely-utilized high performance liquid chromatography methods will be used to measure glycemic control from whole blood samples.
Change from Baseline HbA1c | 6 months
  Widely-utilized high performance liquid chromatography methods will be used to measure glycemic control from whole blood samples.
Change from Baseline HbA1c | 12 months
  Widely-utilized high performance liquid chromatography methods will be used to measure glycemic control from whole blood samples.

SECONDARY OUTCOMES:
Body Mass Index | Baseline
  Calculated measure of body max index from height/weight measures
Change from Baseline Body Mass Index | 3 months
  Calculated measure of body max index from height/weight measures
Change from Baseline Body Mass Index | 6 months
  Calculated measure of body max index from height/weight measures
Change from Baseline Body Mass Index | 12 months
  Calculated measure of body max index from height/weight measures
LDL Cholesterol | Baseline
  Standard enzymatic laboratory procedures will be used to assess total cholesterol, HDL cholesterol, and triglycerides from whole blood. LDL will be calculated based on total cholesterol and HDL values.
Change from baseline LDL Cholesterol | 3 months
  Standard enzymatic laboratory procedures will be used to assess total cholesterol, HDL cholesterol, and triglycerides from whole blood. LDL will be calculated based on total cholesterol and HDL values.
Change from baseline LDL Cholesterol | 6 months
  Standard enzymatic laboratory procedures will be used to assess total cholesterol, HDL cholesterol, and triglycerides from whole blood. LDL will be calculated based on total cholesterol and HDL values.
Change from baseline LDL Cholesterol | 12 months
  Standard enzymatic laboratory procedures will be used to assess total cholesterol, HDL cholesterol, and triglycerides from whole blood. LDL will be calculated based on total cholesterol and HDL values.
Systolic Blood Pressure | Baseline
  A sphygmometer will be assessed to assess systolic blood pressure fifteen minutes after participant is in a seated position with their arm elevated.
Change from baseline Systolic Blood Pressure | 3 months
  A sphygmometer will be assessed to assess systolic blood pressure fifteen minutes after participant is in a seated position with their arm elevated.
Change from baseline Systolic Blood Pressure | 6 months
  A sphygmometer will be assessed to assess systolic blood pressure fifteen minutes after participant is in a seated position with their arm elevated.
Change from baseline Systolic Blood Pressure | 12 months
  A sphygmometer will be assessed to assess systolic blood pressure fifteen minutes after participant is in a seated position with their arm elevated.

OTHER OUTCOMES:
Carbohydrate Management Attitude Scale | Baseline
  Uses a Likert question format (n=12) and assesses attitudes and motivation for carbohydrate management.
Change from baseline Carbohydrate Management Attitude Scale | 3 months
  Uses a Likert question format (n=12) and assesses attitudes and motivation for carbohydrate management.
Change from baseline Carbohydrate Management Attitude Scale | 6 months
  Uses a Likert question format (n=12) and assesses attitudes and motivation for carbohydrate management.
Change from baseline Carbohydrate Management Attitude Scale | 12 months
  Uses a Likert question format (n=12) and assesses attitudes and motivation for carbohydrate management.
Fat Management Attitude Scale | Baseline
  Uses a Likert question format (n=12) and assesses attitudes and motivation for dietary fat management.
Change from baseline Fat Management Attitude Scale | 3 months
  Uses a Likert question format (n=12) and assesses attitudes and motivation for dietary fat management.
Change from baseline Fat Management Attitude Scale | 6 months
  Uses a Likert question format (n=12) and assesses attitudes and motivation for dietary fat management.
Change from baseline Fat Management Attitude Scale | 12 months
  Uses a Likert question format (n=12) and assesses attitudes and motivation for dietary fat management.
Diabetes Empowerment Scale | Baseline
  Uses a Likert question format (n=8) and assesses motivation for overall diabetes self-care.
Change from baseline Diabetes Empowerment Scale | 3 months
  Uses a Likert question format (n=8) and assesses motivation for overall diabetes self-care.
Change from baseline Diabetes Empowerment Scale | 6 months
  Uses a Likert question format (n=8) and assesses motivation for overall diabetes self-care.
Change from baseline Diabetes Empowerment Scale | 12 months
  Uses a Likert question format (n=8) and assesses motivation for overall diabetes self-care.
Problem Areas in Diabetes Scale Questionnaire | Baseline
  Uses a Likert question (n=20) format and assesses patients' problems in applying various self-care areas, including dietary self-care skills.
Change from baseline Problem Areas in Diabetes Scale Questionnaire | 3 months
  Uses a Likert question (n=20) format and assesses patients' problems in applying various self-care areas, including dietary self-care skills.
Change from baseline Problem Areas in Diabetes Scale Questionnaire | 6 months
  Uses a Likert question (n=20) format and assesses patients' problems in applying various self-care areas, including dietary self-care skills.
Change from baseline Problem Areas in Diabetes Scale Questionnaire | 12 months
  Uses a Likert question (n=20) format and assesses patients' problems in applying various self-care areas, including dietary self-care skills.
Situational Obstacles to Dietary Adherence Questionnaire | Baseline
  Uses a Likert question (n=6) format and assesses self-efficacy in adhering to dietary recommendations and managing situations that make adherence challenging (e.g., social activities including few healthy food options.
Change from baseline Situational Obstacles to Dietary Adherence Questionnaire | 3 months
  Uses a Likert question (n=6) format and assesses self-efficacy in adhering to dietary recommendations and managing situations that make adherence challenging (e.g., social activities including few healthy food options.
Change from baseline Situational Obstacles to Dietary Adherence Questionnaire | 6 months
  Uses a Likert question (n=6) format and assesses self-efficacy in adhering to dietary recommendations and managing situations that make adherence challenging (e.g., social activities including few healthy food options.
Change from baseline Situational Obstacles to Dietary Adherence Questionnaire | 12 months
  Uses a Likert question (n=6) format and assesses self-efficacy in adhering to dietary recommendations and managing situations that make adherence challenging (e.g., social activities including few healthy food options.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Matthew Walker Comprehensive Health Center, Nashville, Tennessee
  - Meharry Medical College, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller ST, Akohoue SA, Murry VM, Tabatabai M, Wilus D, Foxx A. SISTER (Sisters Inspiring Sisters to Engage in Relevant Diabetes Self-Care) Diabetes Study: Protocol for diabetes medical nutrition therapy randomized clinical trial among African American women. Contemp Clin Trials. 2023 Feb;125:107052. doi: 10.1016/j.cct.2022.107052. Epub 2022 Dec 13. PMID 36526256